CLINICAL TRIAL: NCT04085575
Title: Efficacy of 1g Versus 2g Intra-auricular Tranexamic Acid in Postoperative Bleeding After Total Knee Arthroplasty
Brief Title: Efficacy of Intra-auricular Tranexamic Acid in Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier de Montauban (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHM
Record Dates: First submitted 2019-08-29; First posted 2019-09-11 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2019-09

CONDITIONS: Postoperative Hemorrhage
MeSH Terms: conditions — Postoperative Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: They were assigned in two groups: The G1 group received 1 g of intra-articular tranexamic acid (TXA) and the G2 group received 2 g of intra-articular tranexamic acid. Both groups received 15 mg / kg IV at 20 min at induction and then 10 mg / kg in oral administration 6 and 12 hours after induction dose IV of tranexamic acid.
Who Masked: Participant, Care Provider
Masking Description: Recruited patients were randomly before the operation by generating random numbers with Microsoft Excel 2007 (Microsoft Corporation, Seattle, Washington, USA).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tranexamic acid - The G1 group (Active Comparator): The G1 group received 1 g of intra-articular tranexamic acid (TXA). The G1 group received 15 mg / kg IV at 20 min at induction and then 10 mg / kg in oral administration 6 and 12 hours after induction dose IV of tranexamic acid.
  Interventions: Drug: Acide Tranexamique
- tranexamic acid - The G2 group (Active Comparator): The G2 group received 2 g of intra-articular tranexamic acid (TXA). The G2 group received 15 mg / kg IV at 20 min at induction and then 10 mg / kg in oral administration 6 and 12 hours after induction dose IV of tranexamic acid.
  Interventions: Drug: Acide Tranexamique

INTERVENTIONS:
Drug: Acide Tranexamique — Recruited patients were randomly before the operation by generating random numbers with Microsoft Excel 2007. They were assigned in two groups: 1 g of intra-articular tranexamic acid (TXA) and 2 g of intra-articular tranexamic acid.
  Other Names: Exacyl

SUMMARY:
Tranexamic acid an antifibrinolytic that develops its anti-haemorrhagic action by inhibiting fibrinolytic activities of plasmin and many studies confirms its effectiveness in decreasing blood loss. The aim of this study was to observe postoperative bleeding with combined intravenous and per - os administration with two intra - articular doses (1 g and 2 g) of tranexamic acid in adult patients undergoing unilateral total knee replacement.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is widely used as an effective treatment for end-stage osteoarthritis and other joint diseases of the knee and it improvements in surgical materials and techniques have greatly increased its effectiveness. However, TKA is an orthopaedic surgical method that has a substantial perioperative blood loss.

Classical methods for reducing blood loss and transfusion rate include the use of a pneumatic tourniquet, intraoperative cell saver, hypotensive anesthesia, application of erythropoietin, autologous blood transfusion, plugging of the femoral canal, cementing, drain clamping, navigation and minimally invasive surgery.

Tranexamic acid (TXA) an antifibrinolytic that develops its anti-haemorrhagic action by inhibiting fibrinolytic activities of plasmin has been used as an adjuvant to such measure and many studies with a level of evidence confirms its effectiveness in decreasing blood loss.

Fibrinolysis is stimulated by surgical trauma blood loss and TKA may be related to increased fibrinolytic activity. TXA inhibits fibrinolysis by blocking the lysine-binding sites of plasminogen to fibrin. Plasmin, bound to tranexamic acid, has a considerably diminished activity with respect to fibrin compared to that of free plasmin. Also, it appears from various studies that, in vivo, tranexamic acid at high doses exerts a braking activity on the activation of the complement system. So, TXA reduces bleeding in the TKA and its functional repercussion has also been confirmed in assays for various dosages and routes of administration.

In the literature, efficacy of intra-articular TXA has also been confirmed, but what is the right dosage is now unclear.

The aim of this study was to observe postoperative bleeding with combined intravenous and per - os administration with two intra - articular doses (1 g and 2 g) of tranexamic acid (Sanofi-Aventis® Gentilly, France).

ELIGIBILITY:
Inclusion Criteria:

- Adult patients undergoing unilateral total knee replacement

Exclusion Criteria:

* Absence of consent
* Tranexamic acid allergy
* Coagulopathy (preoperative platelet count <150,000 / mm3, INR [international normalized ratio]> 1.4, or prolonged partial thromboplastin time> 1.4 times normal),
* History of arterial or venous thromboembolic disease (cerebrovascular accident, deep vein thrombosis or pulmonary thromboembolism),
* Hematological disorder (a hematopoietic, hemorrhagic or thrombogenic disease),
* Retinopathy (severe limitation of the field of vision and / or color distortion),
* Refusal to receive blood products
* Pregnancy
* History of convulsions
* Participation in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2020-01-09 (Actual)

PRIMARY OUTCOMES:
Blood loss in postoperative drainage. | Blood loss in 24 hours postoperative drainage
  The primary endpoint was the bleeding represented by blood loss in postoperative drainage.

SECONDARY OUTCOMES:
The change in hematocrit levels | change in hematocrit levels at 24 and 72 hours
  The secondary outcomes were the change in hematocrit levels.
The change in hemoglobin levels | change in hemoglobin levels at 24 and 72 hours
  The secondary outcomes were the change in hemoglobin levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Edmundo Pereira de Souza Neto, Montauban, Tarn Et Garonne, France

IPD SHARING:
Plan to Share IPD: No
The aim of our study was to observe postoperative bleeding with combined intravenous and per - os administration with two intra - articular doses (1 g and 2 g) of tranexamic acid.

REFERENCES:
- [Derived] Souza Neto EP, Usandizaga G. [Comparison of two doses of intra-articular tranexamic acid on postoperative bleeding in total knee arthroplasty: a randomized clinical trial]. Braz J Anesthesiol. 2020 Jul-Aug;70(4):318-324. doi: 10.1016/j.bjan.2020.03.015. Epub 2020 Jul 8. PMID 32819728